CLINICAL TRIAL: NCT02928393
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Safety, Efficacy and Pharmacodynamic Study of Basmisanil (RO5186582) in Adults With Severe Motor Impairment Following an Ischemic Stroke
Brief Title: A Study to Evaluate the Safety and Efficacy of Basmisanil in Adults With Severe Motor Impairment Following an Ischemic Stroke
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low participant enrolment
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP29937; 2015-003227-66 (EudraCT Number)
Record Dates: First submitted 2016-10-07; First posted 2016-10-10 (Estimated); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Stroke
Keywords: Stroke; Motor impairment; Stroke recovery; Middle cerebral artery stroke; Fugl Meyer; Fugl-Meyer Motor Scale (FMMS)
MeSH Terms: conditions — Stroke; Infarction, Middle Cerebral Artery | interventions — basmisanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Basmisanil (Experimental): Basmisanil at a dose of 240 milligrams (mg) orally twice daily for 90 days.
  Interventions: Drug: Basmisanil
- Placebo (Placebo Comparator): Placebo matched to basmisanil orally twice daily for 90 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Basmisanil — Basmisanil immediate-release granules at a dose of 240 mg will be given orally twice daily for 90 days.
  Other Names: RO5186582
  Arms: Basmisanil
Drug: Placebo — Placebo matched to basmisanil immediate-release granules will be given orally twice daily for 90 days.
  Arms: Placebo

SUMMARY:
This Phase IIa, randomized, double-blind, placebo-controlled, parallel group study will evaluate the safety, efficacy and pharmacodynamics of basmisanil in adult participants with severe motor impairment following an ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Radiologic assessment confirming an acute middle cerebral artery ischemic stroke
* Index stroke occurred within the past 3-4 days
* Inpatient males and females
* Severe hemiparesis or hemiplegia defined by FMMS score less than or equal to (</=) 35
* Sufficient speech, vision and hearing to participate in study evaluations

Exclusion Criteria:

* NIHSS greater than (>) 20
* Severe aphasia that prevents a participant from following directions in rehabilitation
* Significant deficit from prior strokes or pre-existing motor deficit
* History of epilepsy, neurosurgery, severe head trauma or central nervous system infections that have residual symptomatology or have required treatment in the last 12 months
* Known or suspected clinical seizure post-index stroke
* History of pre-existing dementia or use of medications for dementia
* History of clinically significant pre-existing psychiatric conditions within 12 months prior to stroke
* Due to undergo carotid surgery within the next 4 months
* Enrollment/participation in any interventional study (clinical trial) involving an investigational drug (unapproved) or non-drug treatment within the prior 3 months or 6 times the half-life (whichever is longer)
* Clinically relevant medical conditions that would likely interfere with the study conduct and scheduled assessments
* Contraindication to magnetic resonance imaging (MRI) or conditions which render interpretation of MRI difficult

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2017-11-03 (Actual); Study Completion 2017-11-03 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in FMMS Score at Day 90 | Baseline (Day 1), Day 90
Number of Participants with Adverse Events | Baseline (Day 1) up to 28 days after last dose of study drug (latest at Day 118)
Change From Baseline in Montreal Cognitive Assessment (MoCA) Score at Day 30 | Baseline (Day 1), Day 30
Change From Baseline in MoCA Score at Day 90 | Baseline (Day 1), Day 90
Change From Baseline in National Institute of Health Stroke Scale (NIHSS) Score At Day 3 | Baseline (Day 1), Day 3
Change From Baseline in NIHSS Score At Day 10 | Baseline (Day 1), Day 10
Change From Baseline in NIHSS Score At Day 30 | Baseline (Day 1), Day 30
Change From Baseline in NIHSS Score At Day 90 | Baseline (Day 1), Day 90
Change From Baseline in NIHSS Score At 28 Days After Last Dose | Baseline (Day 1) and at 28 days after last dose of study drug (latest on Day 118)
Change From Baseline in Columbia-Suicide Severity Rating Scale (C-SSRS) Score At Day 3 | Baseline (Day 1), Day 3
Change From Baseline in C-SSRS Score At Day 30 | Baseline (Day 1), Day 30
Change From Baseline in C-SSRS Score At Day 60 | Baseline (Day 1), Day 60
Change From Baseline in C-SSRS Score At Day 90 | Baseline (Day 1), Day 90
Change From Baseline in C-SSRS Score At 28 Days After Last Dose | Baseline (Day 1), at 28 days after last dose of study drug (latest on Day 118)

SECONDARY OUTCOMES:
Change From Baseline in Modified Rankin Scale (mRS) Score At Day 90 | Baseline (Day 1), Day 90
mRS Score At Day 90 | Day 90
Change From Baseline in Fugl-Meyer Assessment (FMA) Total Score at Day 90 | Baseline (Day 1), Day 90
Change From Baseline in FMA Subscale Score at Day 90 | Baseline (Day 1), Day 90
Apparent Oral Clearance (CL/F) of Basmisanil | Predose (Hour 0) (prior to morning dose) on Days 3, 10, 30, 90; 4 and 8 hours post-morning dose on Day 1; and 4 hours post-morning dose on Day 3
Maximum Observed Plasma Concentration (Cmax) of Basmisanil | Predose (Hour 0) (prior to morning dose) on Days 3, 10, 30, 90; 4 and 8 hours post-morning dose on Day 1; and 4 hours post-morning dose on Day 3
Apparent Volume of Distribution at Steady States (Vss) of Basmisanil | Predose (Hour 0) (prior to morning dose) on Days 3, 10, 30, 90; 4 and 8 hours post-morning dose on Day 1; and 4 hours post-morning dose on Day 3
Area Under the Curve [AUC] of Basmisanil | Predose (Hour 0) (prior to morning dose) on Days 3, 10, 30, 90; 4 and 8 hours post-morning dose on Day 1; and 4 hours post-morning dose on Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- France (6):
  - CHU de Besancon Hopital Jean Minjoz; Service de Neurologie, Besançon
  - Hôpital Pellegrin Tripode - CHU de Bordeaux, Bordeaux
  - Hopital la Cavale Blanche, Brest
  - Hopital Gabriel Montpied CHU de Clermont-Ferrand; Service de Neurologie B, Clermont-Ferrand
  - Hôpital General - Service de neurologie; Service de neurologie, Dijon
  - Hopital Purpan, Toulouse
- Spain (7):
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital de la Santa Creu i Sant Pau; Servicio de Neurologia, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - La Paz University Hospital, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Virgen del Rocio, Seville
  - Hospital Clnico Universitario de Zaragoza, Zaragoza